CLINICAL TRIAL: NCT03154359
Title: An Open-Label, Single- and Multi-Dose Study to Evaluate the Relationship Between the Pharmacokinetics, Pharmacodynamics, and Clinical Outcomes of Atomoxetine in CYP2D6 Extensive, Intermediate and Poor Metabolizers in Children With Attention Deficit/Hyperactivity Disorder
Brief Title: Atomoxetine PBPK-PD Clinical Study
Status: Completed | Type: Observational
Sponsor: Children's Mercy Hospital Kansas City (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Steve Leeder, Deputy Director, Children's Mercy Research Institute, Children's Mercy Hospital Kansas City
Other Study IDs: 16100728; U54HD090258-01 (NIH)
Record Dates: First submitted 2017-05-04; First posted 2017-05-16 (Actual); Results first posted 2023-08-08 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-08

CONDITIONS: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Atomoxetine Hydrochloride

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Atomoxetine Hydrochloride — Atomoxetine dose adjusted to achieve pre-defined concentration

SUMMARY:
The primary aims of this study focus on characterizing the relationship between atomoxetine exposure and clinical outcomes, as assessed by standardized measures. We will also simultaneously monitor side effect of atomoxetine, another measure of clinical outcomes, and categorize study participants on their ability to tolerate atomoxetine.

DETAILED DESCRIPTION:
Atomoxetine (ATX), Strattera®, is a norepinephrine re-uptake transporter inhibitor that is approved by the Food and Drug Administration (FDA) for the treatment of attention deficit/hyperactivity disorder (ADHD). The drug is often considered a second- or third-line agent, due to the perception that the drug does not work very well. In fact, in a review of studies submitted to the FDA, it reported that there appeared to be discrete classes of response to atomoxetine. After 6-9 weeks of treatment, 47% of the patients were considered "responders" based on changes in the rating scales used to measure ADHD symptoms whereas 40% of patients were considered non-responders. Statistically significant (p<0.001) differences in scores between responders and non-responders were apparent after the first week of treatment. At the relatively low starting doses of the titration scheme, this suggests that there may be a subgroup of patents who are particularly responsive to ATX. We hypothesize that there could be two reasons for this: 1) variability in drug pharmacokinetics (i.e., inadequate drug concentrations in the blood over time could lead to poor response) and 2) variability in drug pharmacodynamics (i.e. differences at the level of the target of drug action that limit the response to a drug, regardless of concentration of drug present in the blood). The CYP2D6 gene, which encodes for the drug metabolizing enzyme CYP2D6, is responsible for the clearance of ATX from the body, is highly polymorphic. ATX metabolism by CYP2D6 protein is one of the major routes of clearance (i.e., removal) of this drug. Genetic variability in the CYP2D6 gene leads to wide inter-individual variability in the activity of the enzyme, ultimately resulting in differing amount of drug in the body (also referred to as "exposure," and is a component of drug pharmacokinetics). Secondly, the SLC6A2 gene which encodes for the norepinephrine reuptake transporter, the drug target for ATX, is also subject to genetic variation. Reported genetic variants of SLC6A2 have been associated with decreased abundance of the transporter. The consequences of SLC6A2 genetic variation with regards to ATX clinical response are currently unknown. In the context of distinct "responder" and "non-responder" groups with a population of atomoxetine-treated patients, non-response could be due to definable differences at the level of the drug target (patients unlikely to respond regardless of the ATX concentrations achieved), or simply a consequence of inadequate exposure in a substantial proportion of population. The goal of this study is to address this issue.

ELIGIBILITY:
Inclusion Criteria:• Males and females 6-18 years of age at the time of enrollment

* Diagnosis of ADHD, as confirmed by a Study Physician at intake visit.
* Intention of the Study Physician to begin therapy with ATX at intake visit
* Willing to provide written permission/assent to participate
* ADHD Medication Status is one of the following:

  * ADHD medication naïve or not currently taking ADHD medication including stimulants, α2-agonists, and ATX, or
  * Currently taking a stimulant for ADHD and is willing to wash out of stimulants prior to starting ATX. This washout is also approved by a Study Physician, or other qualified study personnel (see Section 11.0 for Procedures Involved).

Exclusion Criteria:

* An IQ < 70
* A diagnosis of Autism Spectrum Disorder
* Inability or unwillingness to have blood drawn as described in the protocol schedule of events and consent
* Underlying risk for cardiotoxicity, such as presentation of structural cardiac abnormalities, cardiomyopathy, or arrhythmias
* Clinically significant abnormal safety laboratory values as determined by treating physician
* Diagnosis that may cause abnormal absorption or gastric emptying, such as reflux, inflammatory bowel disease, or Crohn's disease
* For females, a positive urine pregnancy test
* Previous history of adverse drug reaction to ATX
* Use of drugs known to inhibit CYP2D6:

  * Concurrent therapy with sertraline, venlafaxine, imipramine, nortriptyline, quinidine, propafenone, cimetidine, tamoxifen, bupropion, over-the-counter medications containing diphenhydramine, codeine, tramadol, hydrocodone, or oxycodone
  * Concurrent or previous therapy with fluoxetine or paroxetine in the last 2 months
  * Concurrent or previous therapy with terbinafine in the last 6 months
* Unwillingness or inability to washout of stimulant ADHD medications
* Concurrent or recent use of other psychiatric/behavioral health drugs including SSRIs, SNRIs, antipsychotics, anxiolytics, anti-epileptics, and α2-agonists that would impact the participant's pharmacokinetic and/or pharmacodynamic baseline
* Subject is considered by PI to be unsuitable for participation in the study for any reason

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Males and females 6-18 years of age, with a diagnosis of ADHD.
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2017-12-12 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James S Leeder, PharmD, PhD, Principal Investigator — Children's Mercy Hospital Kansas City
Locations (1):
- Children's Mercy Hospital and Clinics, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Newcorn JH, Sutton VK, Weiss MD, Sumner CR. Clinical responses to atomoxetine in attention-deficit/hyperactivity disorder: the Integrated Data Exploratory Analysis (IDEA) study. J Am Acad Child Adolesc Psychiatry. 2009 May;48(5):511-518. doi: 10.1097/CHI.0b013e31819c55b2. PMID 19318988
- [Background] Seneca N, Gulyas B, Varrone A, Schou M, Airaksinen A, Tauscher J, Vandenhende F, Kielbasa W, Farde L, Innis RB, Halldin C. Atomoxetine occupies the norepinephrine transporter in a dose-dependent fashion: a PET study in nonhuman primate brain using (S,S)-[18F]FMeNER-D2. Psychopharmacology (Berl). 2006 Sep;188(1):119-27. doi: 10.1007/s00213-006-0483-3. Epub 2006 Aug 4. PMID 16896954
- [Background] Michelson D, Read HA, Ruff DD, Witcher J, Zhang S, McCracken J. CYP2D6 and clinical response to atomoxetine in children and adolescents with ADHD. J Am Acad Child Adolesc Psychiatry. 2007 Feb;46(2):242-51. doi: 10.1097/01.chi.0000246056.83791.b6. PMID 17242628
- [Background] Kim CH, Hahn MK, Joung Y, Anderson SL, Steele AH, Mazei-Robinson MS, Gizer I, Teicher MH, Cohen BM, Robertson D, Waldman ID, Blakely RD, Kim KS. A polymorphism in the norepinephrine transporter gene alters promoter activity and is associated with attention-deficit hyperactivity disorder. Proc Natl Acad Sci U S A. 2006 Dec 12;103(50):19164-9. doi: 10.1073/pnas.0510836103. Epub 2006 Dec 4. PMID 17146058
- [Background] Gaedigk A, Twist GP, Leeder JS. CYP2D6, SULT1A1 and UGT2B17 copy number variation: quantitative detection by multiplex PCR. Pharmacogenomics. 2012 Jan;13(1):91-111. doi: 10.2217/pgs.11.135. Epub 2011 Nov 23. PMID 22111604
- [Background] Gaedigk A, Simon SD, Pearce RE, Bradford LD, Kennedy MJ, Leeder JS. The CYP2D6 activity score: translating genotype information into a qualitative measure of phenotype. Clin Pharmacol Ther. 2008 Feb;83(2):234-42. doi: 10.1038/sj.clpt.6100406. Epub 2007 Oct 31. PMID 17971818
- [Background] Gaedigk A, Ndjountche L, Divakaran K, Dianne Bradford L, Zineh I, Oberlander TF, Brousseau DC, McCarver DG, Johnson JA, Alander SW, Wayne Riggs K, Steven Leeder J. Cytochrome P4502D6 (CYP2D6) gene locus heterogeneity: characterization of gene duplication events. Clin Pharmacol Ther. 2007 Feb;81(2):242-51. doi: 10.1038/sj.clpt.6100033. PMID 17259947
- [Background] Gaedigk A, Jaime LK, Bertino JS Jr, Berard A, Pratt VM, Bradfordand LD, Leeder JS. Identification of Novel CYP2D7-2D6 Hybrids: Non-Functional and Functional Variants. Front Pharmacol. 2010 Oct 4;1:121. doi: 10.3389/fphar.2010.00121. eCollection 2010. PMID 21833166
- [Background] Gaedigk A, Fuhr U, Johnson C, Berard LA, Bradford D, Leeder JS. CYP2D7-2D6 hybrid tandems: identification of novel CYP2D6 duplication arrangements and implications for phenotype prediction. Pharmacogenomics. 2010 Jan;11(1):43-53. doi: 10.2217/pgs.09.133. PMID 20017671
- [Background] Gaedigk A. Complexities of CYP2D6 gene analysis and interpretation. Int Rev Psychiatry. 2013 Oct;25(5):534-53. doi: 10.3109/09540261.2013.825581. PMID 24151800

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited over 6 years from a patient population seeking care for Attention Deficit Hyperactivity Disorder (ADHD).
Pre-assignment Details: A total of 51 participants were enrolled in the study. All participants completed a screening visit, and 9 participants screenfailed/were determined to be ineligible.
Groups:
- Atomoxetine HCl (Strattera): Study participants will receive atomoxetine at a dose expected to result in steady-state maximum concentration (Cmax,ss) values of 400 ng/mL. Dose will be calculated using a model based on CYP2D6 predicted phenotype, height, weight, body habitus, and gender. Study clinicians may titrate up the dose to reach Cmax,ss values of 600 ng/mL or 800 ng/mL according to participant response.
Period: Overall Study
Arm/Group | Atomoxetine HCl (Strattera)
Started | 42
6 Weeks | 29
18 Weeks | 20
Completed | 20
Not Completed | 22
Not completed — Adverse Event | 1
Not completed — Lack of Efficacy | 2
Not completed — Lost to Follow-up | 3
Not completed — Physician Decision | 3
Not completed — Protocol Violation | 4
Not completed — Withdrawal by Subject | 5
Not completed — Disruption of study due to COVID-19 | 4

BASELINE CHARACTERISTICS:
Groups:
- Atomoxetine HCl (Strattera): Study participants will receive atomoxetine at a dose expected to result in steady-state maximum concentration (Cmax,ss) values of 400 ng/mL. Individualized dose to achieve the desired Cmax,ss of 400 ng/ml (approximately 90 minutes after dose administration) is determined using a pharmacokinetic model that includes as input information each participant's CYP2D6 genotype-predicted phenotype, height, weight, body habitus, and gender. Study clinicians may titrate up the dose to reach predicted Cmax,ss values of 600 ng/mL or 800 ng/mL according to participant response.
Arm/Group | Atomoxetine HCl (Strattera)
Number analyzed (Participants) | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.62 (2.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 40
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 14
  White | 22
  More than one race | 6
  Unknown or Not Reported | 0
Neuropsychiatric Comorbidities [Count of Participants; unit: Participants]
  Anxiety | 3
  Oppositional Defiant Disorder | 4
  Dyslexia | 2
  Learning Delay | 2
  Other | 2
  None | 29
Weight [Mean (Standard Deviation); unit: kilograms (kg)] | 42.93 (20.78)
ADHD Subtype (based on NICHQ Vanderbilt Assessment Scale score) [Count of Participants; unit: Participants] — The NICHQ Vanderbilt Assessment Scales assess the presence and severity of all 18 DSM-V criteria for ADHD (9 inattentive symptoms and 9 hyperactivity/impulsivity symptoms). To meet criteria for an ADHD diagnosis, one must have at least 6 positive responses to the 9 inattentive (inattentive subtype) or 9 hyperactive/impulsivity (hyperactive/impulsive subtype) core symptoms, or both (combined subtype).
  Participants
    Inattentive Subtype | 9
    Hyperactive/Impulsive Subtype | 2
    Combined Subtype | 27
    Below Threshold | 4
ADHD Subtype (based on K-SADS-PL) [Count of Participants; unit: Participants] — The Kiddie Schedule for Affective Disorders and Schizophrenia for School-Age Children - Present and Lifetime Version (K-SADS-PL) is a semi-structured interview that is extensively used in clinical psychology research to diagnose an extensive array of psychopathology, including ADHD and subtype, based on the DSM criteria.
  Participants
    Inattentive Subtype | 16
    Hyperactive/Impulsive Subtype | 3
    Combine Subtype | 21
    Below Threshold | 2
CYP2D6 Activity Score [Count of Participants; unit: Participants] — CYP2D6 genotypes were translated into activity scores as recommended by the Clinical Pharmacogenetics Implementation Consortium (CPIC). Normal function alleles were assigned a value of 1, decreased function alleles a value of 0.25 or 0.5, and non-functional alleles a value of 0; for multiplication events, the value was multiplied by the number of copies detected. The activity score for an individual study participant was assigned as the sum of the scores for each allele, with poor metabolizers defined by an activity score of 0 and ultrarapid metabolizers defined by an activity score >2.25.
  Participants
    0 | 3
    0.25 | 3
    0.5 | 1
    0.75 | 1
    1 | 15
    1.25 | 6
    1.5 | 5
    2 | 7
    3 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Classified as Responders and Non-responders to Intervention
Description: Classification of participants as "responders" versus "non-responders" is based on percent reduction in total National Initiative for Children's Healthcare Quality (NICHQ) Vanderbilt Assessment Scale (3rd edition) score from baseline. Participants with ≥40% reduction in total score from baseline are classified as responders. The scale assesses the presence and severity of 18 DSM-V criteria for attention deficit hyperactivity disorder (ADHD) symptoms. Symptoms are rated on a 4-point Likert-type scale: 0 ("Never") to 3 ("Very Often"). Maximum total symptom score is 54.The measure includes 8 questions assessing functional impairment ("Performance"). Impairment is rated on a 5-point Likert-type scale: 1 ("Excellent") to 5 ("Problematic").
Time Frame: 6 weeks
Population: Individuals who completed 6 week milestone
Measure: Count of Participants; unit: Participants
Groups:
- Atomoxetine HCl (Strattera): Study participants will receive atomoxetine at a dose expected to result in Cmax,ss values of 400 ng/mL. Study clinicians may titrate up the dose to reach Cmax,ss values of 600 ng/mL or 800 ng/mL according to participant response.
Arm/Group | Atomoxetine HCl (Strattera)
Number analyzed (Participants) | 29
Participants
  Responders | 14
  Non-Responders | 15

2. Primary Outcome: Number of Participants Classified as Responders and Non-responders to Intervention
Description: as for outcome 1
Time Frame: 18 weeks
Population: Participants who completed 18 week milestone
Measure: Count of Participants; unit: Participants
Groups:
- Atomoxetine HCl (Strattera): Study participants will receive atomoxetine at a dose expected to result in steady-state maximum concentration (Cmax,ss) values of 400 ng/mL. Study clinicians may titrate up the dose to reach Cmax,ss values of 600 ng/mL or 800 ng/mL according to participant response.
Arm/Group | Atomoxetine HCl (Strattera)
Number analyzed (Participants) | 20
Participants
  Responder | 13
  Non-Responder | 7

3. Primary Outcome: Maximum Plasma Concentration (Cmax) of Atomoxetine
Description: Cmax is the highest concentration of atomoxetine measured over a 12-hour period following administration of the drug on pharmacokinetic study days occurring at baseline (first dose). Cmax is an estimate of atomoxetine systemic exposure and is compared between responders and non-responders.
Time Frame: Baseline (first dose)
Population: 6-week and 18-week responder classifications have different sample sizes, as there are 2 milestones within this study.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Atomoxetine HCl (Strattera)
Number analyzed (Participants) | 29
ng/mL
  Responder at 6 weeks: number analyzed (Participants) | 14
  Responder at 6 weeks | 268.5 (117.2)
  Non-Responder at 6 weeks: number analyzed (Participants) | 15
  Non-Responder at 6 weeks | 220.4 (76.0)
  Responder at 18 weeks: number analyzed (Participants) | 13
  Responder at 18 weeks | 247.8 (128.7)
  Non-Responder at 18 weeks: number analyzed (Participants) | 7
  Non-Responder at 18 weeks | 216.2 (77.3)
Statistical Analysis 1: Comparison: Atomoxetine HCl (Strattera); Comparing 6-week responders and 6-week non-responders; Test type: Other; p = 0.197, t-test, 2 sided
Statistical Analysis 2: Comparison: Atomoxetine HCl (Strattera); Comparing 18-week responders and 18-week non-responders; Test type: Other; p = 0.562, t-test, 2 sided

4. Primary Outcome: Maximum Plasma Concentration (Cmax) of Atomoxetine
Description: Cmax is the highest concentration of atomoxetine measured following administration of the drug on pharmacokinetic study days occurring at 6 weeks. Cmax is an estimate of atomoxetine systemic exposure and is compared between responders and non-responders.
Time Frame: 6 weeks
Population: Participants who completed 6 week milestone
Measure: Mean (Standard Error); unit: ng/mL
Arm/Group | Atomoxetine HCl (Strattera)
Number analyzed (Participants) | 29
ng/mL
  Responders: number analyzed (Participants) | 14
  Responders | 554.2 (63.5)
  Non-Responders: number analyzed (Participants) | 15
  Non-Responders | 501.7 (61.4)
Statistical Analysis 1: Comparison: Atomoxetine HCl (Strattera); Test type: Other; p = 0.558, t-test, 2 sided

5. Primary Outcome: Maximum Plasma Concentration (Cmax) of Atomoxetine
Description: Cmax is the highest concentration of atomoxetine measured following administration of the drug on pharmacokinetic study days occurring at 18 weeks. Cmax is an estimate of atomoxetine systemic exposure and is compared between responders and non-responders.
Time Frame: 18 weeks
Population: The overall participants were classified into 2 groups based on responder status.
Measure: Mean (Standard Error); unit: ng/mL
Arm/Group | Atomoxetine HCl (Strattera)
Number analyzed (Participants) | 20
ng/mL
  Responders: number analyzed (Participants) | 13
  Responders | 601.3 (88.2)
  Non-Responders: number analyzed (Participants) | 7
  Non-Responders | 375.5 (120.2)
Statistical Analysis 1: Comparison: Atomoxetine HCl (Strattera); Test type: Other; p = 0.147, t-test, 2 sided

6. Primary Outcome: Area Under the Plasma Concentration-time Curve (AUC) of Atomoxetine
Description: AUC is the area under the plasma concentration-time curve following administration of atomoxetine. For the baseline pharmacokinetic study (first dose of atomoxetine) plasma concentrations were measured at 17 timepoints between 0 and 72 hours (0, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16, 20, 24, 48, and 72 hours) post-dose for CYP2D6 poor and intermediate metabolizers, and 12 timepoints between 0 and 12 hours (0, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, and 12 hours) after dose administration for all other participants. The AUC was generated using a mixed log-linear approach and extrapolated to infinity. AUC is compared between responders and non-responders.
Time Frame: Baseline (first dose)
Population: 6-week and 18-week responder classifications have different sample sizes, as there are 2 milestones within this study.
Measure: Mean (Standard Deviation); unit: (ng*hours)/mL
Arm/Group | Atomoxetine HCl (Strattera)
Number analyzed (Participants) | 29
(ng*hours)/mL
  Responder at 6 weeks: number analyzed (Participants) | 14
  Responder at 6 weeks | 1515.3 (1169.2)
  Non-responder at 6 weeks: number analyzed (Participants) | 15
  Non-responder at 6 weeks | 1246.9 (913.4)
  Responder at 18 weeks: number analyzed (Participants) | 13
  Responder at 18 weeks | 1495.7 (1197.6)
  Non-responder at 18 weeks: number analyzed (Participants) | 7
  Non-responder at 18 weeks | 1462.7 (1283.4)
Statistical Analysis 1: Comparison: Atomoxetine HCl (Strattera); Comparing 6-week responders and 6-week non-responders; Test type: Other; p = 0.495, t-test, 2 sided
Statistical Analysis 2: Comparison: Atomoxetine HCl (Strattera); Comparing 18-week responders and 18-week non-responders; Test type: Other; p = 0.955, t-test, 2 sided

7. Primary Outcome: Area Under the Plasma Concentration-time Curve (AUC) of Atomoxetine
Description: For the steady-state pharmacokinetic studies at 6 weeks, plasma concentrations were measured at 15 timepoints between 0 and 24 hours (0, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16, 20, and 24 hours) post-dose for CYP2D6 poor and intermediate metabolizers, and at 12 timepoints between 0 and 12 hours (0, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, and 12 hours) and extrapolated to 24 hours for all other participants. AUC is compared between responders and non-responders.
Time Frame: 6 weeks
Population: The overall participants were classified into 2 groups based on responder status.
Measure: Mean (Standard Error); unit: (ng*hours)/mL
Arm/Group | Atomoxetine HCl (Strattera)
Number analyzed (Participants) | 29
(ng*hours)/mL
  Responders: number analyzed (Participants) | 14
  Responders | 2802.5 (423.4)
  Non-Responders: number analyzed (Participants) | 15
  Non-Responders | 2809.4 (409.0)
Statistical Analysis 1: Comparison: Atomoxetine HCl (Strattera); Test type: Other; p = 0.991, t-test, 2 sided

8. Primary Outcome: Area Under the Plasma Concentration-time Curve (AUC) of Atomoxetine
Description: For the steady-state pharmacokinetic studies at 18 weeks, plasma concentrations were measured at 15 timepoints between 0 and 24 hours (0, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16, 20, and 24 hours) post-dose for CYP2D6 poor and intermediate metabolizers, and at 12 timepoints between 0 and 12 hours (0, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, and 12 hours) and extrapolated to 24 hours for all other participants. AUC is compared between responders and non-responders.
Time Frame: 18 weeks
Population: The overall participants were classified into 2 groups based on responder status.
Measure: Mean (Standard Error); unit: (ng*hours)/mL
Arm/Group | Atomoxetine HCl (Strattera)
Number analyzed (Participants) | 20
(ng*hours)/mL
  Responders: number analyzed (Participants) | 13
  Responders | 3149.2 (511.3)
  Non-Responders: number analyzed (Participants) | 7
  Non-Responders | 2880.0 (696.7)
Statistical Analysis 1: Comparison: Atomoxetine HCl (Strattera); Test type: Other; p = 0.759, t-test, 2 sided

9. Primary Outcome: Plasma Concentration of 3,4-dihydroxyphenylglycol (DHPG)
Description: DHPG has been proposed as a biomarker of the activity of the norepinephrine reuptake transporter (NET; SLC6A2), the target of atomoxetine action. DHPG is a degradation product of norepinephrine after it has been taken up by pre-synaptic neurons, and higher concentrations in plasma are considered to reflect higher NET activity (higher reuptake of norepinephrine into pre-synaptic neurons). To assess the potential value of DHPG as a biomarker of atomoxetine response in ADHD, absolute baseline and pre-dose concentrations of DHPG will be compared between atomoxetine responders and non-responders.
Time Frame: Baseline
Population: 6-week and 18-week responder classifications have different sample sizes, as there are 2 milestones within this study.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Atomoxetine HCl (Strattera)
Number analyzed (Participants) | 29
ng/mL
  Responder at 6 weeks: number analyzed (Participants) | 14
  Responder at 6 weeks | 0.363 (0.164)
  Non-responder at 6 weeks: number analyzed (Participants) | 15
  Non-responder at 6 weeks | 0.412 (0.178)
  Responder at 18 weeks: number analyzed (Participants) | 13
  Responder at 18 weeks | 0.382 (0.177)
  Non-responder at 18 weeks: number analyzed (Participants) | 7
  Non-responder at 18 weeks | 0.363 (0.184)
Statistical Analysis 1: Comparison: Atomoxetine HCl (Strattera); Comparing 6-week responders and 6-week non-responders; Test type: Other; p = 0.456, t-test, 2 sided
Statistical Analysis 2: Comparison: Atomoxetine HCl (Strattera); Comparing 18-week responders and 18-week non-responders; Test type: Other; p = 0.822, t-test, 2 sided

10. Primary Outcome: Plasma Concentration of 3,4-dihydroxyphenylglycol (DHPG)
Description: DHPG has been proposed as a biomarker of the activity of the norepinephrine reuptake transporter (NET; SLC6A2), the target of atomoxetine action. DHPG is a degradation product of norepinephrine after it has been taken up by pre-synaptic neurons, and higher concentrations in plasma are considered to reflect higher NET activity (higher reuptake of norepinephrine into pre-synaptic neurons). To assess the potential value of DHPG as a biomarker of atomoxetine response in ADHD, pre-dose concentration of DHPG at the 6-week pharmacokinetic study visit will be compared between atomoxetine responders and non-responders.
Time Frame: 6 weeks
Population: The overall participants were classified into 2 groups based on responder status.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Atomoxetine HCl (Strattera)
Number analyzed (Participants) | 29
ng/mL
  Responders: number analyzed (Participants) | 14
  Responders | 0.395 (0.150)
  Non-Responders: number analyzed (Participants) | 15
  Non-Responders | 0.345 (0.125)
Statistical Analysis 1: Comparison: Atomoxetine HCl (Strattera); Test type: Other; p = 0.343, t-test, 2 sided

11. Primary Outcome: Plasma Concentration of 3,4-dihydroxyphenylglycol (DHPG)
Description: DHPG has been proposed as a biomarker of the activity of the norepinephrine reuptake transporter (NET; SLC6A2), the target of atomoxetine action. DHPG is a degradation product of norepinephrine after it has been taken up by pre-synaptic neurons, and higher concentrations in plasma are considered to reflect higher NET activity (higher reuptake of norepinephrine into pre-synaptic neurons). To assess the potential value of DHPG as a biomarker of atomoxetine response in ADHD, pre-dose concentration of DHPG at the 18-week pharmacokinetic study visit will be compared between atomoxetine responders and non-responders.
Time Frame: 18 weeks
Population: The overall participants were classified into 2 groups based on responder status.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Atomoxetine HCl (Strattera)
Number analyzed (Participants) | 20
ng/mL
  Responders: number analyzed (Participants) | 13
  Responders | 0.323 (0.140)
  Non-responders: number analyzed (Participants) | 7
  Non-responders | 0.283 (0.139)
Statistical Analysis 1: Comparison: Atomoxetine HCl (Strattera); Test type: Other; p = 0.539, t-test, 2 sided

12. Primary Outcome: Change in Plasma Concentration of DHPG From Baseline
Description: The change in DHPG will be compared between atomoxetine responders and non-responders.
Time Frame: 6 weeks
Population: The overall participants were classified into 2 groups based on responder status.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Atomoxetine HCl (Strattera)
Number analyzed (Participants) | 29
ng/mL
  Responders: number analyzed (Participants) | 14
  Responders | 0.031 (0.180)
  Non-Responders: number analyzed (Participants) | 15
  Non-Responders | -0.066 (0.157)
Statistical Analysis 1: Comparison: Atomoxetine HCl (Strattera); Test type: Other; p = 0.130, t-test, 2 sided

13. Primary Outcome: Change in Plasma Concentration of DHPG From Baseline
Description: The change in DHPG will be compared between atomoxetine responders and non-responders.
Time Frame: 18 weeks
Population: The overall participants were classified into 2 groups based on responder status.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Atomoxetine HCl (Strattera)
Number analyzed (Participants) | 20
ng/mL
  Responders: number analyzed (Participants) | 13
  Responders | -0.059 (0.074)
  Non-responders: number analyzed (Participants) | 7
  Non-responders | -0.081 (0.140)
Statistical Analysis 1: Comparison: Atomoxetine HCl (Strattera); Test type: Other; p = 0.652, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over the full 18 weeks of participation in the study.
Arm/Group | Atomoxetine HCl (Strattera)
All-Cause Mortality (participants affected / at risk) | 0/42
Serious Adverse Events (participants affected / at risk) | 0/42
Other Adverse Events (participants affected / at risk) | 37/42
OTHER ADVERSE EVENTS (reported when occurring in more than 2.5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Atomoxetine HCl (Strattera) (N=42)
Nausea/Vomiting/Upset Stomach (Gastrointestinal disorders) | 20
Decreased Appetite (Gastrointestinal disorders) | 4
Diarrhea (Gastrointestinal disorders) | 2
Cold/Flu (Infections and infestations) | 10
Fever (Infections and infestations) | 2
Ear Infection (Infections and infestations) | 2
Sore Throat (Infections and infestations) | 2
Headache (Nervous system disorders) | 9
Irritability (Psychiatric disorders) | 2
Mood Disturbance (Psychiatric disorders) | 2
Self-Injurious Behavior (Psychiatric disorders) | 2
Fatigue (General disorders) | 8
Foot injury (Musculoskeletal and connective tissue disorders) | 2

LIMITATIONS AND CAVEATS:
Recruitment was severely affected by the COVID-19 pandemic, and did not recover as hospital operations adapted to the pandemic. Therefore, study was terminated before enrollment goal was met.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-04-01): https://cdn.clinicaltrials.gov/large-docs/59/NCT03154359/Prot_SAP_000.pdf